CLINICAL TRIAL: NCT05000879
Title: A Randomized Controlled Trial of Mental Health Outcomes and Putative Targets of an Online Mindfulness Program for New and Expectant Mothers
Brief Title: How Does Mindful Mood Balance for Moms Work?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, CHRISTINA METCALF, Senior Instructor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-0402
Record Dates: First submitted 2021-08-05; First posted 2021-08-11 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Depression; Pregnancy Related; Antenatal Depression; Depression, Postpartum
MeSH Terms: conditions — Depression; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMB for Moms (Experimental): Subjects will receive digital delivery of Mindful Mood Balance for Moms for 12 weeks. Subjects will be unconstrained in the types of treatments or other wellness activities they could receive while participating in the study.
  Interventions: Behavioral: MMB for Moms
- Waitlist Control (No Intervention): Subjects will be unconstrained in the types of treatments or other wellness activities they could receive while participating in the study.

INTERVENTIONS:
Behavioral: MMB for Moms — 12-week program that emphasizes mindfulness and cognitive behavioral skills
  Arms: MMB for Moms

SUMMARY:
The purpose of this investigation is to conduct a randomized trial comparing a web-based Mindful Mood Balance for Moms course without coaching support to waitlist control among pregnant or early parenting women with depression histories.

DETAILED DESCRIPTION:
Mindfulness-based cognitive therapy (MBCT) prevents depressive relapse and reduces residual depression symptoms among adults with recurrent depression not currently in episode. Women in perinatal or early parenting years constitute a significant portion of this at-risk population with a history of depression for whom MBCT was designed. Novel delivery formats that provide access to core knowledge and skills of MBCT could increase public health impact-particularly for perinatal or early parenting women-but it is unclear whether such formats have comparable mental health outcomes and changes in putative targets as in-person MBCT.

In the present study, we planned to randomize 60 pregnant or early parenting women with a history of major depression and current residual depressive symptoms to MMB for Moms, a web-based course that teaches skills from MBCT customized specifically for pregnant and postpartum women, or waitlist control. We planned to address the following specific aims:

Aim 1. We evaluated the extent to MMB for Moms was associated with significant reduction in residual depression symptoms as compared to WLC. We predicted the rate of change in depression symptoms across the study would be greater on average for participants randomized to MMB for Moms relative to those randomized to WLC.

Aim 2. We evaluated the extent to MMB for Moms significantly engaged the putative target of decentering as compared to WLC. We predicted the rate of change in decentering across the study would be greater on average for participants randomized to MMB for Moms relative to participants randomized to WLC.

Aim 3. We evaluated the extent to MMB for Moms significantly engaged the putative target of self-compassion as compared to WLC. We predicted the rate of change in self-compassion across the study would be greater on average for participants randomized to MMB for Moms relative to participants randomized to WLC.

ELIGIBILITY:
Inclusion Criteria:

1. female,
2. pregnant or having had a child within the past 36 months, *
3. 18 years of age or older,
4. having a history of one or more prior major depressive episode (as assessed by a single question, "Have you had a history of mood concerns or major depression?")
5. a current PHQ-9 score of <= 14, and
6. endorses ability to read and write fluently in English.

Exclusion Criteria:

1. meeting criteria for current moderately severe depression symptoms (as assessed by the PHQ-9 >= 15),
2. current imminent suicidality (as assessed by the PHQ-9), and
3. indication of other disorders or symptoms that necessitate priority treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Rate of change in depression symptoms | Through 6-month follow-up
  Change in the severity of depressive symptoms will be evaluated by the Patient Health Questionnaire-9 (PHQ-9)
Rate of change in decentering | Through 6-month follow-up
  Change in decentering will be evaluated by the Experiences Questionnaire-Decentering subscale
Rate of change in self-compassion | Through 6-month follow-up
  Change in self-compassion will be evaluated by the Self-Compassion Scale (SCS)
Depressive Relapse Status | Through 6-month follow-up
  Rate of depressive relapse will be assessed using the Lifetime Depression Assessment Self-report (LIDAS), adapted to reference the past 3 or 6 months based on survey completion.
Rate of change in anxiety symptoms | Through 6-month follow-up
  Change in the severity of anxiety symptoms will be evaluated by the 3. Generalized Anxiety Disorder-7 (GAD-7)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and accompanying documentation will be available for use by other investigators upon request.
Time Frame: Data will become available after study completion.
Access Criteria: Interested investigators will be asked to submit a proposal form, which will be reviewed by the principal investigators for scientific integrity and adherence to ethical guidelines.

REFERENCES:
- [Background] Dimidjian S, Goodman SH, Felder JN, Gallop R, Brown AP, Beck A. Staying well during pregnancy and the postpartum: A pilot randomized trial of mindfulness-based cognitive therapy for the prevention of depressive relapse/recurrence. J Consult Clin Psychol. 2016 Feb;84(2):134-45. doi: 10.1037/ccp0000068. Epub 2015 Dec 14. PMID 26654212